CLINICAL TRIAL: NCT03540706
Title: Impact of the Use of C-reactive Protein in a Micro-method on the Prescription of Antibiotics in General Practitioners Consulting in the Office
Brief Title: Impact of the Use of CRP on the Prescription of Antibiotics in General Practitioners
Acronym: VIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: VIP; 2018-A00242-53 (Other: ID-RCB); AOR17072 (Other Grant/Funding Number: GIRCI IDF)
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Respiratory Infection; Respiratory Infections in Children
Keywords: Respiratory Infections; C-reactive protein; antibiotic prescription
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care with C-reactive protein assay in micro method (Experimental): During a visit to the general practitioner for a clinical suspicion of respiratory infection, the doctor will practice a C-reactive protein assay in micro method. He will prescribe antibiotics according to the result of the dosage
  Interventions: Diagnostic Test: Care with C-reactive protein assay in micro method
- Care without C-reactive protein assay in micro method (No Intervention): Simple management of a patient coming for a suspicion of respiratory infection without dosage of the C-reactive protein in micro method

INTERVENTIONS:
Diagnostic Test: Care with C-reactive protein assay in micro method — Care with C-reactive protein assay in micro method
  Arms: Care with C-reactive protein assay in micro method

SUMMARY:
Respiratory infections, including episodes of coughing with fever, are the main cause of outpatient antibiotic prescription, while a minority of them are linked to bacterial infections requiring antibiotic. These prescriptions are often performed by general practitioners. These unnecessary antibiotic contribute to increased bacterial resistance, side effects and unnecessary costs. Campaigns for the correct prescription of antibiotics have had a real but partial or transient success.

C-reactive protein micro-method (POCT-CRP) could help to differentiate between viral and bacterial infections and thus contribute to the proper use of antibiotics. The decrease in prescription of antibiotics is likely to have an even stronger positive impact in countries like France, where prescription is high.

The objective of this study is to evaluate the use of POCT-CRP in the general practitioner's office in case of suspected respiratory infection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 3 years
* Clinical suspicion of respiratory infection defined by the presence of at least one respiratory sign among, cough, dyspnea, chest pain and auscultatory abnormality and at least one general sign among fever, sweat, headache, myalgia, impairment of general condition
* Affiliated to a social health insurance
* Signed consent

Exclusion Criteria:

* Duration of symptoms < 24 hours
* Hospitalization or emergency assessment decision decided from the outset
* Signs of severity before the realization of POCT-CRP
* Patient previously included in the study for the same episode
* Antibiotic therapy within 7 days
* Chronic cough (more than 3 weeks)

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Frequency of antibiotic therapy prescribed | 10 days
  with and without POCT-CRP

SECONDARY OUTCOMES:
Frequency of antibiotic therapy prescribed in patients aged from 3 to 17 years old | 10 days
  with and without POCT-CRP
Frequency of antibiotic therapy prescribed in patients aged from 18 to 64 years old | 10 days
  with and without POCT-CRP
Frequency of antibiotic therapy prescribed in patients older than 65 years old | 10 days
  with and without POCT-CRP
Type of antibiotic prescribed | 10 days
Frequency of complementary exam | 10 days
  with and without POCT-CRP
type of complementary exam | 10 days
  with and without POCT-CRP
Proportion of number of patients referred to emergency | 10 days
  with and without POCT-CRP
Proportion of number of patients with delayed antibiotic therapy | 10 days
  with and without POCT-CRP
number of prescription following the recommended algorythms | 10 days
  Adequacy between the proposed decision algorithm according to the C-reactive protein assay and the antibiotic prescription
Concordance between the prescription proposed by the decision algorithm as a function of the micro-CRP and the prescription realized: kappa coefficient | 10 days
  The assessment of the utility of the POCT procedure
COVID-19 positive patients | 1 day
  Number of COVID-19 positive patients by diagnostic method (From October 2020)

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - 22 rue de Silly, Boulogne
  - 18 rue Sainte Bathilde, Chelles
  - 25 avenue des frères Lumière, Cormeilles-en-Parisis
  - 8 Rue Saint-Exupéry, Meudon-la-Forêt
  - 258 Bis Rue de Paris, Montreuil
  - 61bis Boulevard de Charonne, Paris
  - 25 Rue de Fécamp, Paris
  - 237 Rue de la Croix Nivert,, Paris
  - 1 Rue Colette Magny, Paris
  - 391 Rue des Pyrénées, Paris
  - 50 Rue de la Justice, Paris
  - 72 Boulevard Davout, Paris
  - 20 avenue Gorges Sand, Stains
  - 19 Rue du Midi, Vincennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gulliford MC, Moore MV, Little P, Hay AD, Fox R, Prevost AT, Juszczyk D, Charlton J, Ashworth M. Safety of reduced antibiotic prescribing for self limiting respiratory tract infections in primary care: cohort study using electronic health records. BMJ. 2016 Jul 4;354:i3410. doi: 10.1136/bmj.i3410. PMID 27378578
- [Background] Llor C, Moragas A, Cots JM, Lopez-Valcarcel BG; Happy Audit Study Group. Estimated saving of antibiotics in pharyngitis and lower respiratory tract infections if general practitioners used rapid tests and followed guidelines. Aten Primaria. 2017 Jun-Jul;49(6):319-325. doi: 10.1016/j.aprim.2016.07.002. Epub 2016 Nov 22. PMID 27884552
- [Background] van Vugt SF, Verheij TJ, de Jong PA, Butler CC, Hood K, Coenen S, Goossens H, Little P, Broekhuizen BD; GRACE Project Group. Diagnosing pneumonia in patients with acute cough: clinical judgment compared to chest radiography. Eur Respir J. 2013 Oct;42(4):1076-82. doi: 10.1183/09031936.00111012. Epub 2013 Jan 24. PMID 23349450
- [Background] Huang Y, Chen R, Wu T, Wei X, Guo A. Association between point-of-care CRP testing and antibiotic prescribing in respiratory tract infections: a systematic review and meta-analysis of primary care studies. Br J Gen Pract. 2013 Nov;63(616):e787-94. doi: 10.3399/bjgp13X674477. PMID 24267862
- [Background] Kapasi AJ, Dittrich S, Gonzalez IJ, Rodwell TC. Host Biomarkers for Distinguishing Bacterial from Non-Bacterial Causes of Acute Febrile Illness: A Comprehensive Review. PLoS One. 2016 Aug 3;11(8):e0160278. doi: 10.1371/journal.pone.0160278. eCollection 2016. PMID 27486746
- [Background] Ivaska L, Niemela J, Leino P, Mertsola J, Peltola V. Accuracy and feasibility of point-of-care white blood cell count and C-reactive protein measurements at the pediatric emergency department. PLoS One. 2015 Jun 2;10(6):e0129920. doi: 10.1371/journal.pone.0129920. eCollection 2015. PMID 26034987
- [Background] Esposito S, Tremolati E, Begliatti E, Bosis S, Gualtieri L, Principi N. Evaluation of a rapid bedside test for the quantitative determination of C-reactive protein. Clin Chem Lab Med. 2005;43(4):438-40. doi: 10.1515/CCLM.2005.077. PMID 15899661
- [Background] Cohen R, Lecuyer A, Wollner C, Deberdt P, Thollot F, Henriquet V, de La Rocque F. [Evaluation of impact of CRP rapid test in management of febrile children in ambulatory pediatric practice]. Arch Pediatr. 2008 Jun;15(6):1126-32. doi: 10.1016/j.arcped.2008.03.007. Epub 2008 May 16. French. PMID 18486458
- [Background] Cohen R, Romain O, Levy C, Perreaux F, Decobert M, Hau I, Lecuyer A, Lesprit E, Maman L, Roullaud S, Cheron G, Bekri A, d'Athis P, Henriquet V, de La Rocque F. [Impact of CRP rapid test in management of febrile children in paediatric emergency units of Ile-de-France]. Arch Pediatr. 2006 Dec;13(12):1566-71. doi: 10.1016/j.arcped.2006.09.003. Epub 2006 Oct 27. French. PMID 17070024
- [Background] Do NT, Ta NT, Tran NT, Than HM, Vu BT, Hoang LB, van Doorn HR, Vu DT, Cals JW, Chandna A, Lubell Y, Nadjm B, Thwaites G, Wolbers M, Nguyen KV, Wertheim HF. Point-of-care C-reactive protein testing to reduce inappropriate use of antibiotics for non-severe acute respiratory infections in Vietnamese primary health care: a randomised controlled trial. Lancet Glob Health. 2016 Sep;4(9):e633-41. doi: 10.1016/S2214-109X(16)30142-5. Epub 2016 Aug 3. PMID 27495137
- [Background] Minnaard MC, van de Pol AC, Hopstaken RM, van Delft S, Broekhuizen BD, Verheij TJ, de Wit NJ. C-reactive protein point-of-care testing and associated antibiotic prescribing. Fam Pract. 2016 Aug;33(4):408-13. doi: 10.1093/fampra/cmw039. Epub 2016 May 26. PMID 27230745
- [Background] Verlee L, Verheij TJ, Hopstaken RM, Prins JM, Salome PL, Bindels PJ. [Summary of NHG practice guideline 'Acute cough']. Ned Tijdschr Geneeskd. 2012;156(0):A4188. Dutch. PMID 22917039
- [Background] van Vugt SF, Broekhuizen BD, Lammens C, Zuithoff NP, de Jong PA, Coenen S, Ieven M, Butler CC, Goossens H, Little P, Verheij TJ; GRACE consortium. Use of serum C reactive protein and procalcitonin concentrations in addition to symptoms and signs to predict pneumonia in patients presenting to primary care with acute cough: diagnostic study. BMJ. 2013 Apr 30;346:f2450. doi: 10.1136/bmj.f2450. PMID 23633005
- [Background] Cals JW, Hopstaken RM, Butler CC, Hood K, Severens JL, Dinant GJ. Improving management of patients with acute cough by C-reactive protein point of care testing and communication training (IMPAC3T): study protocol of a cluster randomised controlled trial. BMC Fam Pract. 2007 Mar 29;8:15. doi: 10.1186/1471-2296-8-15. PMID 17394651
- [Background] Little P, Stuart B, Francis N, Douglas E, Tonkin-Crine S, Anthierens S, Cals JW, Melbye H, Santer M, Moore M, Coenen S, Butler C, Hood K, Kelly M, Godycki-Cwirko M, Mierzecki A, Torres A, Llor C, Davies M, Mullee M, O'Reilly G, van der Velden A, Geraghty AW, Goossens H, Verheij T, Yardley L; GRACE consortium. Effects of internet-based training on antibiotic prescribing rates for acute respiratory-tract infections: a multinational, cluster, randomised, factorial, controlled trial. Lancet. 2013 Oct 5;382(9899):1175-82. doi: 10.1016/S0140-6736(13)60994-0. Epub 2013 Jul 31. PMID 23915885
- [Background] Marrie TJ, Durant H, Yates L. Community-acquired pneumonia requiring hospitalization: 5-year prospective study. Rev Infect Dis. 1989 Jul-Aug;11(4):586-99. doi: 10.1093/clinids/11.4.586. PMID 2772465
- [Background] Prina E, Ranzani OT, Torres A. Community-acquired pneumonia. Lancet. 2015 Sep 12;386(9998):1097-108. doi: 10.1016/S0140-6736(15)60733-4. Epub 2015 Aug 12. PMID 26277247
- [Background] Houck PM, Bratzler DW, Nsa W, Ma A, Bartlett JG. Timing of antibiotic administration and outcomes for Medicare patients hospitalized with community-acquired pneumonia. Arch Intern Med. 2004 Mar 22;164(6):637-44. doi: 10.1001/archinte.164.6.637. PMID 15037492
- [Background] Meehan TP, Fine MJ, Krumholz HM, Scinto JD, Galusha DH, Mockalis JT, Weber GF, Petrillo MK, Houck PM, Fine JM. Quality of care, process, and outcomes in elderly patients with pneumonia. JAMA. 1997 Dec 17;278(23):2080-4. PMID 9403422
- [Background] Colvin JM, Muenzer JT, Jaffe DM, Smason A, Deych E, Shannon WD, Arens MQ, Buller RS, Lee WM, Weinstock EJ, Weinstock GM, Storch GA. Detection of viruses in young children with fever without an apparent source. Pediatrics. 2012 Dec;130(6):e1455-62. doi: 10.1542/peds.2012-1391. Epub 2012 Nov 5. PMID 23129086
- [Background] Hernandez-Bou S, Trenchs V, Vanegas MI, Valls AF, Luaces C. Evaluation of the bedside Quikread go(R) CRP test in the management of febrile infants at the emergency department. Eur J Clin Microbiol Infect Dis. 2017 Jul;36(7):1205-1211. doi: 10.1007/s10096-017-2910-2. Epub 2017 Feb 3. PMID 28160147
- [Background] Llor C, Bjerrum L, Munck A, Cots JM, Hernandez S, Moragas A; HAPPY AUDIT Investigators. Access to point-of-care tests reduces the prescription of antibiotics among antibiotic-requesting subjects with respiratory tract infections. Respir Care. 2014 Dec;59(12):1918-23. doi: 10.4187/respcare.03275. PMID 25468986